CLINICAL TRIAL: NCT03144661
Title: A Phase 1, Open-Label, Dose-Escalation and Expansion, Safety and Tolerability Study of INCB062079 in Subjects With Advanced Hepatocellular Carcinoma and Other Malignancies
Brief Title: An Open-Label Safety and Tolerability Study of INCB062079 in Subjects With Advanced Hepatocellular Carcinoma and Other Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Strategic Business Decision
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INCB 62079-101; 2017-001153-13 (EudraCT Number)
Record Dates: First submitted 2017-05-05; First posted 2017-05-09 (Actual); Last update posted 2025-10-21 (Actual); Status verified 2025-10

CONDITIONS: Hepatocellular Carcinoma (HCC); Cholangiocarcinoma; Esophageal Cancer; Nasopharyngeal Cancer; Ovarian Cancer; Solid Tumors
Keywords: hepatocellular carcinoma; cholangiocarcinoma; esophageal; nasopharyngeal; serous ovarian; solid tumors; fibroblast growth factor (FGF); fibroblast growth factor receptor (FGFR)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Cholangiocarcinoma; Esophageal Neoplasms; Nasopharyngeal Neoplasms; Ovarian Neoplasms; Acrocephalosyndactylia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Part 1 - INCB062079 10mg QD (Experimental): INCB062079 was administered at 10mg once daily
  Interventions: Drug: INCB062079
- Part 1 - INCB062079 10mg BID (Experimental): NCB062079 was administered at 10mg twice daily
  Interventions: Drug: INCB062079
- Part 1 - INCB062079 15mg BID (Experimental): NCB062079 was administered at 15mg twice daily
  Interventions: Drug: INCB062079
- Part 1 - INCB062079 10 mg BID + BAS (Experimental): NCB062079 was administered at 10 mg twice daily in combination with bile acid sequestrants (BAS)
  Interventions: Drug: INCB062079
- Part 1 - INCB062079 15 mg BID + BAS (Experimental): NCB062079 was administered at 15mg twice daily in combination with bile acid sequestrants (BAS)
  Interventions: Drug: INCB062079
- Part 2 Dose Expansion - Cohort A (Experimental): HCC Subjects with FGF19 amplification were enrolled to evaluate the dose selected in Part 1
  Interventions: Drug: INCB062079
- Part 2 - Dose Expansion Cohort B (Experimental): HCC Subjects without FGF19 amplification were enrolled to evaluate the dose selected in Part 1
  Interventions: Drug: INCB062079
- Part 2 - Dose Expansion Cohort C (Experimental): Subjects with cholangiocarcinoma or esophageal, nasopharyngeal, or serous ovarian cancers (regardless of FGF/FGFR status), or other solid tumor malignancies with documented FGF19/FGFR4 alteration were enrolled to evaluate the dose selected in Part 1
  Interventions: Drug: INCB062079

INTERVENTIONS:
Drug: INCB062079 — In Part 1, initial cohort dose of INCB062079 at the protocol-defined starting dose, with subsequent dose escalations based on protocol-specific criteria. The recommended dose(s) from Part 1 will be taken forward into Part 2 cohorts.

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability, and determine the maximum tolerated dose of INCB062079 in subjects with advanced hepatocellular carcinoma and other malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Part 1: HCC; cholangiocarcinoma; or esophageal, nasopharyngeal, or serious ovarian cancer, regardless of FGF19/FGFR4 status; or other solid tumor malignancies with documented FGF19/FGFR4 alteration (FGF19/FGFR4 pathway activating alterations include, but are not limited to, FGFR4 amplification, FGFR4 activating mutations, and FGF19 amplification) based on local testing.
* Part 2: Subjects will be enrolled into 1 of 3 cohorts:

  * Cohort A: HCC with FGF19 amplification.
  * Cohort B: HCC without FGF19 amplification.
  * Cohort C: cholangiocarcinoma, esophageal, nasopharyngeal or serous ovarian cancers (regardless of FGF19/FGFR4 status), or other solid tumor malignancies with documented FGF19/FGFR4 alteration.
* Has progressed after prior therapy and either a) there is no further effective standard anticancer therapy available (including subject refusal) or b) is intolerant to standard anticancer therapy.
* Life expectancy > 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1 (Part 1) or 0-2 (Part 2).
* Archival tumor specimen according to protocol-defined criteria.
* Centrally analyzed screening C4 (bile acid synthesis precursor) results must be below 40.9 ng/mL, which is the upper limit as determined by the sponsor.
* Must agree to take bile acid sequestrants while taking INCB062079.

Exclusion Criteria:

* Treatment with other investigational study drug for any indication for any reason, or receipt of anticancer medications within 28 days before first dose of study drug; subjects must have recovered from AEs due to previously administered therapies.
* Prior receipt of a selective FGFR4 inhibitor within the last 6 months.
* Laboratory parameters outside the protocol-defined ranges.
* History or presence of an abnormal ECG that in the investigator's opinion is clinically meaningful.
* Prior radiotherapy within 2 weeks of study treatment. A 1-week washout period is permitted for palliative radiation to non- central nervous system (CNS) disease with medical monitor approval.
* History of human immunodeficiency virus infection.
* Untreated brain or CNS metastases or brain/CNS metastases that have progressed. Subjects with previously treated and clinically stable brain/CNS metastases and who are off all corticosteroids for ≥ 4 weeks are eligible.
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment, except concomitant antiviral systemic therapy for chronic hepatitis B or C.
* Child-Pugh liver function Class B or C.
* History of clinically significant or uncontrolled cardiac disease.
* History of allergic reactions to INCB062079, any of the excipients of INCB062079 or similar compounds.
* Pregnant or nursing women or subjects expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 90 days after last dose of study drug.
* Any medical condition that would in the investigator's judgment interfere with full participation in the study, including administration of study medication and attending required study visits; pose a significant risk to the subject; or interfere with interpretation of study data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2020-06-10 (Actual); Study Completion 2020-06-10 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of INCB062079 as measured by assessment of adverse events (AEs) | Baseline to 30-35 days after end of treatment, up to approximately 6 months per subject.
  An AE is defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related, that occurs after a subject provides informed consent.

SECONDARY OUTCOMES:
Objective Response Rate | Every 2 cycles during the treatment period and every 8 weeks during the follow-up period, up to approximately 6 months per subject.
  Defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per modified Response Evaluation Criteria (RECIST) in hepatocellular carcinoma (HCC) and standard Response Evaluation Criteria (RECIST v1.1) in participants with other advanced malignancies.
Cmax of INCB062079 | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject.
  Defined as maximum observed plasma concentration.
Tmax of INCB062079 | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject.
  Defined as time to maximum plasma concentration.
Cmin of INCB062079 | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject.
  Defined as minimum observed plasma concentration during the dosing interval.
AUC0-t of INCB062079 | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject.
  Defined as area under the single-dose plasma concentration-time curve from Hour 0 to the last quantifiable measurable plasma concentration.
t½ of INCB062079 | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject.
  Defined as the apparent plasma terminal phase disposition half-life.
Cl/F of INCB062079 | Protocol-defined time points during Cycles 1 and 2 of treatment, up to approximately 2 months per subject.
  Defined as oral dose clearance.
Analysis of biomarkers | Screening visit
  A plasma sample will be collected during screening for possible analysis of FGFR4 pathway mutations using tumor circulating DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Luis F. Vinas, MD, Study Director — Incyte Corporation
Locations (6):
- United States (3):
  - University of Alabama, Birmingham, Alabama
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Toledo Medical Center, Toledo, Ohio
- Belgium (3):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - University Hospital (UZ) Leuven, Leuven

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Harding JJ, Jungels C, Machiels JP, Smith DC, Walker C, Ji T, Jiang P, Li X, Asatiani E, Van Cutsem E, Abou-Alfa GK. First-in-Human Study of INCB062079, a Fibroblast Growth Factor Receptor 4 Inhibitor, in Patients with Advanced Solid Tumors. Target Oncol. 2023 Mar;18(2):181-193. doi: 10.1007/s11523-023-00948-8. Epub 2023 Feb 14. PMID 36787089